CLINICAL TRIAL: NCT06515964
Title: Development and Validation of a Curability Evaluation Model for Endoscopic Resection of Early Esophageal Squamous Cell Carcinoma Based on China Early Esophageal Cancer Cohort
Brief Title: China Early Esophageal Cancer Cohort
Status: Recruiting | Type: Observational
Sponsor: Changhai Hospital (Other)
Collaborators: Lianshui People's Hospital (Unknown); The second affiliated hospital of Xuzhou medical university (Unknown); The second people's hospital of Nanyang (Unknown); Nanchong Central Hospital (Other Government); Tongliao City Hospital (Unknown); Yancheng First People's Hospital (Other); The Second Hospital of Hebei Medical University (Other); The Second Affiliated Hospital of Baotou Medical College (Other); Affiliated Hospital of Southwest Medical University (Other); Sichuan Cancer Hospital and Research Institute (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Zhongda Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); West China Hospital (Other); The First Affiliated Hospital of Soochow University (Other); Jiangsu Province Hospital of Traditional Chinese Medicine (Other); Shandong Provincial Hospital (Other Government); Shanxi Provincial People's Hospital (Other Government); Henan Provincial People's Hospital (Other); Anyang Cancer Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: CEEC
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Early Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational study — observational study, no intervention

SUMMARY:
With the development of endoscopy, more and more patients with superficial esophageal squamous cell carcinoma (ESCC) receive endoscopic resection rather than traditional surgery. However, there is still no complete consensus on the risk factors for lymph node metastasis (LNM) and recurrence of ESCC after endoscopic resection. The existing curative resection criteria are strict to a certain extent, and a considerable number of patients are overtreated according to the current standard of additional treatment. Thus, we aim to conduct a multi-center retrospective and prospective study to construct a large cohort of ESCC based on the previously established multi-center collaborative research network and clinical big data, analyze the risk factors of LNM and recurrence in patients with early esophageal squamous cell carcinoma after ESD, establish an accurate and simple risk prediction model, and evaluate the discrimination efficiency of this model.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged 18-85.
2. ESD was performed for early (superficial) esophageal squamous cell carcinoma, and the indication was in line with domestic and foreign guidelines.
3. The pathological stage after ESD was pT1a/pT1b.
4. The effective follow-up time after ESD was ≥3 years, or recurrence or LNM occurred during the follow-up period.

Exclusion Criteria:

1. Esophageal chemoradiotherapy or esophageal surgery were performed before ESD.
2. There is a history of carcinoma, early carcinoma, adenoma and other benign and malignant tumors of stomach and duodenum.
3. Pathological data after ESD were incomplete.
4. Combined with malignant tumors of other organs.
5. Fragmented endoscopic mucosal resection (EMR), multi-loop mucosal resection (MBM) and other endoscopic non-monolithic resection techniques were used.
6. New squamous cell carcinoma in other parts of esophagus during follow-up (metachronous carcinoma).

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From January 2015 to December 2020, no less than 1400 patients who received ESD treatment for early esophageal squamous cell carcinoma were expected to be included.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Noncurative Resection | 2022-12 Complete the preliminary clinical study preparation. 2023-10 Complete patient data analysis and sorting. 2024-10 Construct an accurate evaluation system. 2025-10 Conduct validation analysis of the evaluation system.
  Noncurative resection was defined as the presence of residual tumor or lymph node metastasis at the vertical margin of the lesion confirmed by pathology after surgery, or local recurrence, lymph node metastasis, or distant metastasis attributable to the primary tumor during follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No